CLINICAL TRIAL: NCT03030586
Title: A Multi-centre Proof-of-performance Clinical Study to Validate Blood-based Biomarker Candidates for the Diagnosis of Alzheimer's Disease
Brief Title: ADDIA Proof-of-Performance Clinical Study
Acronym: ADDIA
Status: Completed | Type: Observational
Sponsor: Amoneta Diagnostics SAS (Industry)
Collaborators: European Commission (Other); Firalis SA (Industry); University Hospital, Strasbourg (Other); Centre Hospitalier Universitaire Vaudois (Other); IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other); Hopitaux Civils de Colmar (Other); Istanbul University (Other); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Lille (Other); University Hospital, Geneva (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Erasme University Hospital (Other); University Hospital, Montpellier (Other); Centre Hospitalier Universitaire de Besancon (Other); Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: ST0056
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease (AD); Frontotemporal Lobar Degeneration; Dementia with Lewy Bodies (DLB); Parkinson Disease Dementia (PDD); Progressive Supranuclear Palsy (PSP); Corticobasal Degeneration (CBD)
Keywords: Blood cell biomarkers, peripheral circulating biomarkers
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Lobar Degeneration; Lewy Body Disease; Supranuclear Palsy, Progressive; Corticobasal Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Alzheimer: 400 patients in total, with approximately 200 patients with mild Alzheimer's disease and 200 patients with moderate to severe Alzheimer's disease will be recruited for sampling blood, urine (and other peripheral body fluids: tears and saliva as optional) for validation of biomarkers
  Interventions: Other: volumetric MRI
- Non-Alzheimer neurodegenerative disease: 200 patients comprising:
  * 75 patients with behavioural variant of Fronto-Temporal Lobe Degeneration (FTD),
  * 50 patients with Parkinson's disease dementia (PDD),
  * 50 patients with Dementia with Lewy Bodies (DLB) and
  * 25 patients with Progressive Supranuclear Palsy (PSP) or cortico-basal degeneration (CBD)
  Interventions: Other: volumetric MRI
- Healthy Controls: 200 healthy subjects
  Interventions: Other: volumetric MRI

INTERVENTIONS:
Other: volumetric MRI

SUMMARY:
The objective of the ADDIA clinical Proof-of-Performance study is to validate the performance of ADDIA' blood biomarkers for diagnosis of Alzheimer's disease (AD).

ADDIA clinical study is a multi-centre, non-interventional, prospective, proof-of-performance study with only one visit.

About 800 well-characterized subjects will be recruited into 3 groups in 2:1:1 ratio, namely patients with Alzheimer's disease (AD), patients with non-AD neurodegenerative disease (NAD) and 200 control subjects (healthy as compared to their age).

* 400 patients with Alzheimer's disease (AD): 200 patients with mild AD, 200 patients with moderate-to-severe AD,
* 200 patients with non-Alzheimer's neurodegenerative diseases (NAD),
* 200 controls (healthy as compared to their age).

DETAILED DESCRIPTION:
ADDIA study is dedicated to the proof-of-performance (PoP) of blood biomarkers for diagnosis of Alzheimer's disease (AD) and will recruit approximately 800 subjects (400 AD and 400 non-AD).

CONTEXT OF USE:

To quantify the performance of ADDIA' blood biomarkers for AD diagnosis (yes/no).

Since the main objective of this study is to establish the performance of ADDIA' blood cell-based biomarkers β-amyloid (Aβ) and protein kinase C (PKC) and corresponding assays and to seek approval as In-Vitro Diagnosis (IVD) test(s) specific for diagnosis of AD, and to validate the newly identified metabolomics and RNA signatures and selected protein biomarker candidates, samples will be used from:

* the patients recruited in the AD group and patients recruited in the non-AD neurodegenerative disorders (NAD) group who are accurately diagnosed during the pre-screening period, including by using three types of diagnostic methods: clinical neuropsychological scores, neuroimaging (at least volumetric structural MRI) and retrospective cerebrospinal (CSF) data: Aβ, total-Tau and p-tau biomarkers. Alternatively to absence of retrospective CSF data, retrospective Aβ PET /Tau PET scans can be used if compatible to diagnosis of respective diseases.
* the subjects recruited in the control group have no objective memory loss, normal results on neuropsychology tests, and normal neuroimaging findings for their age, as well as normal Aβ PET scan Tau PET scan and normal CSF Aβ, total-Tau and p-Tau concentration if retrospectively available.

For further validation of ADDIA' biomarkers, an integrative tool combining ADDIA' blood biomarkers with cognitive scores and/or, neuroimaging (and/or retrospective CSF biomarker data) will be used. The impact of polymorphisms associated with AD, such as APOE e4 (known to be as risk factor of AD) on ADDIA' blood biomarkers will also be studied.

OBJECTIVES:

Objective 1: Validate the ADDIA biomarker candidates: two blood cell-based biomarkers measured by flow cytometry using Amoneta Diagnostics' proprietary probes specific to beta-Amyloid (Aβ) peptide and protein kinase C (PKC).

ADDIA' blood cell-based Aβ and/or PKC biomarkers will also be combined via an integrative tool with clinical neuropsychological scores (MMSE, MoCA, FCSRT) and/or neuroimaging (at least volumetric MRI) scores for diagnosis and/or differential diagnosis. The impact on these ADDIA biomarkers of genotyping in particular polymorphisms known to be associated with AD (e.g. APOE e4, e2 alleles) will also be tested. In addition, the levels of ADDIA' blood cell-based Aβ and/or PKC biomarkers will be correlated to the levels of CSF biomarkers Aβ and tau or phospho-tau (or Aβ PET and TAU PET levels).

Objective 2: ADDIA clinical PoP study will also validate additional new biomarker candidates (identified previously and/or under analytical validation in the ADKIT study and chronobiological studies) for AD diagnosis in peripheral body fluids; in particular, studies on a set of proteins (using immuno-detection methods), metabolomics/lipidomics signatures (using e.g. LC-HRMS method) and miRNA signature (using e.g. qPCR, HTG-NGS methods) are planned. These new biomarkers may be used if needed to further enhance the accuracy of ADDIA' blood-based Aβ and PKC biomarker test for diagnosis or differential diagnosis.

STUDY DESIGN

ADDIA clinical study is a multi-centre, non-interventional, prospective, proof-of-performance group study without a clinical follow-up. About 800 well characterized subjects will be enrolled into 3 groups in 2:1:1 ratio, namely Alzheimer's disease, non-AD neurodegenerative diseases and controls (healthy as compared to their age). The number of subjects is divided into 3 groups as following:

* 400 patients with Alzheimer's disease (AD),
* 200 patients with non-Alzheimer's neurodegenerative diseases (NAD),
* 200 controls (CC).

All groups will be age-matched and mean age similar in the three groups.

ADDIA clinical study needs to recruit well characterized subjects in each group, therefore a pre-screening or a diagnostic workup of the subjects needs to be performed by the clinical centres before the start of the clinical study (during Visit 0). In ADDIA clinical study, only one visit (Visit 1) is required for the subjects without any follow-up, in which the subjects will be recruited and sampling of blood and urine will be done in the same Visit 1. The following data sets will be collected:

1. Data set 1 and samples available from visit 0 collected in the e-CRF after informed consent signature:

   • Data from all subjects of the three groups include neuropsychological scores (MMSE, MoCA, FCSRT scores), neuroimaging (at least structural MRI volumetric scores, and other neuroimaging as needed for diagnosis) and laboratory data (haematology, biochemistry) related to pre-screening and diagnosis. CSF samples obtained retrospectively by clinical centres are needed if available.
2. Data set 2 and samples from Visit 1 include in all three groups clinical MMSE, FCSRT, MoCA tests (MMSE and MoCA tests to be redone on Visit 1 if older than 3 months) and laboratory data (haematology, biochemistry), and blood and urine (and saliva and tear as optional) collected during Visit 1 (clinical centres). The clinical centres equipped with flow cytometry can perform experiments on ADDIA blood cell-based biomarkers utilizing Amoneta' proprietary Aβ and PKC probes.

Data set 3 will be obtained at the end of ADDIA clinical study (Amoneta Diagnostics/Firalis) and will comprise data on the performance of ADDIA biomarkers as described in details in objectives 1, 2.

SUBJECT RECRUITMENT AND SAMPLING

The subjects who meet the inclusion and exclusion criteria prior to the inclusion in the study (as checked by the clinical centres during Visit 0) will be enrolled in the ADDIA study after the informed consent signatures. Sampling will be performed for the following body fluids during Visit 1: blood (11 tubes, 2.5, 4 or 5 mL each) and urine (1 tube, 5 mL) from all subjects. Saliva (1 tube, 4 mL) and tear (2 tubes, 0.15 mL each) samples are optional.

Eleven tubes of blood and spot urine will be collected from each subject that has fasted for > 12 hours. The samples will be used as follows:

* 2 (two) tubes will be used at the participating clinical centres for routine lab tests, haematology and biochemistry.
* 9 (nine) tubes will be sent to Amoneta facilities in the following format:
* 3 (three) fresh whole blood samples (3 Li-heparin tubes), 1 tube will be sent in the morning immediately after sampling to the flow cytometry laboratory (Amoneta laboratories or another laboratory chosen by Amoneta which can be a laboratory of the clinical centre if equipped with flow cytometry platform) to quantify the performance of ADDIA assays based on blood cell-based biomarkers Aβ and PKC for AD diagnosis and 2 tubes will be used to fix or prepare cells that will be later analysed by flow cytometry at Amoneta laboratories.
* 6 (six) fresh blood samples will be prepared on-site to obtain serum (dry tube), plasma (EDTA and Li-Heparin tubes), PAXgene and PAXRNA samples and PBMC (Li-Heparin tube) samples, which will be aliquoted and stored immediately at -80°C at the clinical centres before being shipped at -80°C later on Amoneta/Firalis central laboratory for testing: genotyping and gene, RNA expression (2 blood tubes), protein expression and metabolomics/lipidomics (1 Li-Heparin and 1 EDTA tubes of plasma, 1 dry tube of serum, and 1 Li-Heparin tube of PBMCs) during the ADDIA program and for validating the emerging biomarkers and for replication studies during or after the ADDIA program (as may be requested by regulatory authorities for IVD product approval).
* Urine samples (and saliva, tear samples as optional) will be aliquoted and frozen immediately at -80°C at the clinical centres and shipped at -80°C to Amoneta/Firalis central laboratory for testing in selected assays based on results that will be obtained on blood samples.

ENDPOINTS

* Performance evaluation of the ADDIA blood biomarkers Aβ and PKC (IVD) kit by AD diagnosis in the form of binary outcome (Yes/No) after quantification of sensitivity & specificity of these biomarkers. This will be also achieved by using the integrative tool enabling comparison of ADDIA blood-based biomarkers Aβ and PKC to and combination with standard clinical diagnosis tests: cognitive scores, neuroimaging scores (and CSF Biomarkers if possible).
* Performance evaluation of the ADDIA' additional new biomarkers (RNA signature, metabolomics signature and/or other peripheral biomarkers) for AD diagnosis in the form of binary outcome (Yes/No) after quantification of sensitivity & specificity of these biomarkers.

STATISTICAL CONSIDERATIONS

Primary consideration (for the evaluation of the diagnostic performance) will be the comparisons between the following groups:

* AD (Mild AD + Moderate-to-severe AD) versus healthy controls, and/or
* Mild AD versus healthy controls, and/or
* Moderate-to-severe AD versus healthy controls, and/or
* AD versus healthy controls+NAD groups.

Secondary considerations (for the evaluation of the differential diagnostic performance) will be the comparisons between the following groups:

* AD (Mild AD + Moderate-to-severe AD) versus NAD and/or
* Mild AD versus NAD and/or
* Moderate-to-severe AD versus NAD and/or
* Mild AD versus Moderate-to-severe AD Tertiary considerations will explore potential differences between NAD versus healthy controls and the subgroups of NAD (FTD, LBD, PDD, PSP, CBD) two by two as well as versus healthy controls and AD.

ELIGIBILITY:
Inclusion Criteria:

For all groups:

* Female and male subjects aged 40 to 85 years.
* Dated and signed informed consent by the subject (or its legal representative if applicable in accordance with the local regulations).
* AD, NAD patients and control subjects will be age-matched and mean age similar in the three groups.
* Able to comply with all study procedures.

For AD group:

* Diagnosis of AD: typical and atypical AD.
* MMSE score (measured in the last 3 months): < 21 for patients with moderate to severe AD. MMSE score > 21 in subjects with mild AD with sporadic or a familial form of AD due to mutation in APP or PSEN1 or PSEN2 genes.
* FCSRT, MoCA tests (MoCA measured in the last 3 months).
* Neuroimaging compatible with a diagnosis of AD:

  * At least quantitative volumetric structural MRI: volumes of hippocampus and cortical areas.
  * Visual semi-quantitative MRI if practiced shall show medial temporal lobe atrophy (MTA) and parietal atrophy with visual rating (semi-quantitative) on the MTA-score (e.g. Scheltens' scores 0-4). MTA score must be ≥ 2 in patients aged 40-75 years and ≥ 3 in patients aged above 75 years. For patients younger than 60 years, and with familial form of AD, who may have normal MTA-scores, Koedam score (0-3) for Parietal Atrophy showing atrophy of the precuneus characteristic of AD may be used with a Koedam score from 1 to 3.

Other neuroimaging data (retrospectively available) including PET Amyloid scan and FDG PET are desired if practiced by clinical centres and if available.

- Cerebrospinal fluid biomarker data (retrospectively available) showing positive levels of at least 2 out of 3 biomarkers: i.e. Aβ1-42 and tau (phosphorylated-Tau and/or total-Tau). Note: If retrospective CSF data are not available, retrospective Aβ PET and Tau PET data can be used.

For NAD group:

For all patients of the group NAD, except PSP subgroup (when PSP has a clear-cut typical phenotype, sometimes called Steele-Richardson phenotype), the CSF biomarker data must show levels for CSF biomarkers Aβ1-42, phosphorylated-Tau and total-Tau, compatible with the respective NAD subgroup. If retrospective CSF data are not available, retrospective Aβ PET and Tau PET data can be used.

Fronto-temporal dementia (FTD)

* Diagnosis of probable behavioural FTD (bvFTD) for all subjects of this FTD subgroup, whether with familial or non-familial forms. If with familial form, the subject must be a member of family with a known mutation in one of the FTD related genes: MAPT, PGRN. The predominant phenotype in the kindred must be cognitive/behavioural (i.e. kindred in whom Parkinsonism or Amyotrophic Lateral Sclerosis is the predominant clinical phenotype among affected relatives is excluded).
* Centrally rated frontal and/or anterior temporal atrophy score of 2 or greater on brain MRI.
* MMSE score compatible. If currently taking an acetylcholinesterase inhibitor and/or memantine, the subject must have been taking such medication(s) for ≥3 months.

Dementia Lewy body (DLB)

* DLB should be diagnosed when dementia occurs before or concurrently with Parkinsonism.
* Patients diagnosed with probable DLB. Probable DLB can be made with the presence of two core features out of the following:

  * Fluctuating cognition with pronounced variations in attention and alertness,
  * Recurrent visual hallucinations that are typically well formed and detailed,
  * Spontaneous features of Parkinsonism.

Probable DLB is diagnosed with the presence of one or more of the above core features and one or more of the following suggestive features. Probable DLB should not be diagnosed on the basis of suggestive features alone:

* REM sleep behaviour disorder,
* Severe neuroleptic sensitivity,
* Low dopamine transporter uptake in basal ganglia demonstrated by SPECT or PET imaging (if data retrospectively available).

Supportive diagnosis:

* Generalized low uptake on SPECT/PET perfusion scan with reduced occipital activity (if data retrospectively available),
* Abnormal (low uptake) MIBG myocardial scintigraphy,
* Prominent slow wave activity on EEG with temporal lobe transient sharp waves.

  * MRI: Relative preservation of medial temporal lobe structures on CT/MRI scan.
  * Clinical Dementia Rating (CDR) score is greater than or equal to 0.5.
  * MMSE score compatible.
  * Patients with familial forms caused by mutation in genes SNCA, SNCB.

Parkinson's disease dementia (PDD)

* Subjects with Parkinson's Disease Dementia (PDD) must have dementia after (not before) developing Parkinson's disease (PD).
* PD is diagnosed by the 3 typical PD symptomatic findings:

  * tremor,
  * rigidity, and
  * slowed movement (bradykinesia).
* Subjects with dementia and with LRRK2 gene mutation (or with mutation in one of the following genes: PARK2 or SNCA, VPS35, PINK1, DJ1, ATP13A2, FBX07, SLC6A3, TAF1 are also included.
* L-DOPA responsive (a good response to levodopa as practiced by clinical investigator, retrospectively to the study).
* MMSE score < 21 for moderate to severe PDD and > 21 for mild PDD.
* MRI: evidence of relevant structural abnormality (i.e. basal ganglia for Parkinsonism and potentially medio-temporal or cortical findings that may be related to dementia). Functional imaging techniques such as fluoro-dopa PET, FDG PET or SPECT to document the presence of dopaminergic dysfunction if retrospectively available.

Progressive Supranuclear Palsy (PSP)

* Diagnosis of probable or possible PSP as defined by the National Institute of Neurological Disorders and Stroke and Society for Progressive Supranuclear Palsy (NINDS-SPSP) diagnostic criteria, and as summarized by Armstrong et al. (2013) for the conclusions on CBD criteria from an international consortium of behavioural neurology, neuropsychology, and movement disorders specialists):

  * Gradually progressive disorder,
  * Onset at age 40 or later,
  * Vertical (upward or downward gaze) supranuclear palsy and prominent postural instability with tendency to fall in the first year of disease onset,
  * No evidence of other diseases that could explain the foregoing features, as indicated by mandatory exclusion criteria.
* Brain MRI at Screening consistent with PSP: neuroradiologic evidence of relevant structural abnormality in the midbrain and frontal lobes (i.e. basal ganglia, lobar atrophy).
* MMSE score compatible.
* Be able to ambulate and stand unassisted for 5 minutes.
* Be able to cooperate with gait and balance testing.

Corticobasal degeneration (CBD)

• Diagnosis of possible CBD. Inclusion clinical criteria for possible CBD, with features of Cortico-Basal Syndrome (CBS); familial forms related to MAPT included, Progressive Supranuclear Palsy Syndrome (PSPS) phenotype included.

* Features of CBS: a) limb rigidity or akinesia, b) limb dystonia, c) limb myoclonus plus 1 of: d) orobuccal or limb apraxia, e) cortical sensory deficit, f) alien limb phenomena (more than simple levitation).
* Features of PSPS: Three of: a) axial or symmetric limb rigidity or akinesia, b) postural instability or falls, c) urinary incontinence, d) behavioural changes, e) supranuclear vertical gaze palsy or decreased velocity of vertical saccades.

Note: subjects with probable sporadic CBD (no familial form) are excluded.

* MRI findings: parietal cortical atrophy (asymmetric).
* MMSE score compatible.

Controls

* Normal cognitive performance with normal scores of neuropsychological tests for their age.
* MMSE >26 (performed in less than 3 months).
* At least volumetric structural MRI with normal findings. Normal retrospective finding in β-amyloid PET scan, FDG PET scan if practiced by clinical centres.
* If retrospectively available, normal CSF biomarkers concentrations: negative levels for all three CSF biomarkers Aβ1-42, phosphorylated-Tau and total-Tau.
* If retrospectively available, Aβ PET and/or Tau PET scan(s) shall be negative.
* Able to comply with the study procedures.

EXCLUSION CRITERIA for all subjects:

The following exclusion criteria apply to all subjects:

* Neutropenia (Neutrophils: < 1,500/mm3 according to ethnic group).
* Thrombocytopenia (platelets: < 100,000/mm3, rule out EDTA-induced pseudo-thrombocytopenia).
* Subjects with less than an elementary education are excluded.
* Subject with no medical insurance are excluded in the countries where medical insurance is mandatory such as in France. In the countries where medical insurance is not mandatory, subjects with no medical insurance may not be excluded.
* Psychiatric history: schizophrenia, psychosis.
* Vascular dementia.
* Infection diseases, chronic inflammatory diseases that affect blood cells, patients with an active infection/ immunosuppressive disorders/ treatment with immunosuppressive or immunomodulatory medication.
* Current malignancy or past diagnosis of malignancy affecting blood cells under treatment or with treatment stopped only during last 3 months.
* Medication interfering with cognitive functions and ADDIA biomarkers (i.e. kinase inhibitors and beta-amyloid and tau passive and active immunizations).
* Major sensory deficits that could interfere with cognitive assessment (visual and auditory).
* Epilepsy.
* Patients with known contraindication for MRI imaging such as MRI-incompatible stent or MRI-incompatible endoprosthesis.

EXCLUSION CRITERIA for AD group

* Mixed dementia.
* Vascular dementia.
* Other dementia type.
* Other neurodegenerative disease.
* Absence of CSF biomarker data and/or amyloid PET data is an exclusive criterion for all subjects with sporadic forms of AD, but it is not an exclusive criterion for subjects with a familial form of AD that is due to a mutation of a gene among APP, PSEN1, PSEN2.

EXCLUSION CRITERIA for NAD group

* AD diagnosis.
* Mixed dementia.
* Vascular dementia.
* Absence of either CSF biomarker data or amyloid PET data is an exclusive criterion for all subjects in sporadic DLB, PDD, FTD and CBD (but not for subjects with PSP when PSP has a clear-cut typical phenotype, sometimes called Steele-Richardson phenotype). However, absence of CSF biomarker and/or amyloid PET data is not an exclusive criterion for subjects with a familial form of NAD that is due to a mutation of a gene among MAPT, PGRN, SNCA, SNCB, PARK2 or SNCA, VPS35, PINK1, DJ1, ATP13A2, FBX07, SLC6A3 or TAF1, TREM2.

EXCLUSION CRITERIA for Control group

* AD patients.
* Dementia patients.
* Cognitive impairments.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: About 800 well characterized subjects will be enrolled into 3 groups in 2:1:1 ratio, namely patients with Alzheimer's disease (AD), patients with non-AD neurodegenerative disease (NAD) and control subjects (healthy as compared to their age). The number of subjects is divided into 3 groups as following:
  * 400 patients with AD (50% with mild AD and 50% of with moderate to severe AD),
  * 200 patients with non-Alzheimer's neurodegenerative diseases (NAD): this group will comprise 75 patients with behavioural variant of Fronto-Temporal Lobe Degeneration (FTD) recruited according to Rascovsky et al., 2011; 50 patients with Parkinson's disease dementia (PDD), 50 patients with Lewy Body dementia (DLB) recruited according to McKeith et al., 2005 criteria; 25 patients with Progressive Supranuclear Palsy (PSP) or cortico-basal degeneration (CBD).
  * 200 controls (healthy as compared to their age).
Sampling Method: Non-Probability Sample
Enrollment: 821 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Blood cell biomarkers for diagnosis of Alzheimer | 18 Months
  Proof of Performance of ADDIA' blood biomarker-based test

SECONDARY OUTCOMES:
Biomarkers circulating in body fluids for diagnosis of Alzheimer and/or other dementia type | 18 months
  Validation of biomarkers circulating in peripheral body fluids

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Blanc, MD, Principal Investigator — Hôpitaux Universitaires Strasbourg; Jean-François Démonet, MD, Principal Investigator — Centre hospitalier universitaire vaudois, Lausanne; Hakan Gurvit, MD, Principal Investigator — Istanbul University, Istanbul; Moira Marizzoni, PhD, Principal Investigator — IRCCS Centro San Giovanni di Dio Fatenenefratelli, Bressia; François Sellal, MD, Principal Investigator — Hôpitaux Civils (Hopital Louis Pasteur) de Colmar; Frisoni Giovanni, MD, Principal Investigator — University Hospital, Geneva; Florence Pasquier, MD, Principal Investigator — Centre Hospitalier Régional, Universitaire de Lille; Adrian Ivanoiu, MD, Principal Investigator — Cliniques Universitaires Saint-Luc, Brussels; Bruno Dubois, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Jean-Christophe Bier, MD, Principal Investigator — Hopital ERASME, Brussels; Audrey Gabelle, MD, Principal Investigator — University Hospital, Montpellier; Eloi Magnin, MD, Principal Investigator — Centre Hospitalier Universitaire de Besançon; Renaud David, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (13):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - ERASME Hospital, Brussels
- France (7):
  - Hopitaux Universitaires de Strasbourg, Strasbourg, Alsace
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Hôpitaux Civils (Hopital Louis Pasteur) de Colmar, Colmar
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nice, Nice
  - APHP-Hôpitaux Universitaires Pitié Salpêtrière, Paris
- IRCCS Centro San Giovanni di Dio Fatenenefratelli, Brescia, Brescia, Italy
- Switzerland (2):
  - Hôpitaux Universitaires de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- Istanbul University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No